CLINICAL TRIAL: NCT00753350
Title: An Open-label, Single-center, Feasibility Study Designed to Evaluate the Safety and Tolerability of Sensate™ Anchored Gastric Device in Subjects With Non-morbid Obesity
Brief Title: METHOD (Minimally Invasive, Endoscopically-delivered, Tolerable by Human Individuals, Non-morbid Obesity Device) Study
Acronym: SENSATE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sensate LLC (Industry)
Collaborators: Johannes Gutenberg University Mainz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SN-101-MZ
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Obesity, Non-morbid
Keywords: obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Sensate™ anti-Obesity device
  Interventions: Device: Sensate™ anchored gastric device

INTERVENTIONS:
Device: Sensate™ anchored gastric device — Delivery/anchoring of the Sensate™ device in the stomach. Withdrawal of the Sensate™ device and its anchoring components after 8 weeks.

SUMMARY:
This will be an open label, single-center, feasibility study comprised of two sequential cohorts( cohort 1: 2 participants; cohort 2: 8 participants).

This study will be conducted in generally healthy participants aged 25 to 55 years with non-morbid obesity and a pre-screening body mass index between 35 and 40.

Participants will undergo screening to determine their health status and their eligibility to participate in the study. Eligible patients will undergo an endoscopic device delivery procedure during which the device will be anchored in the inner stomach wall at the distal anterior antrum. Physical examination and/or endoscopic safety evaluations will be conducted on day 14 and 28. The device and its anchor will be completely removed endoscopically after 8 weeks. The participants will be followed-up for safety evaluation for an additional period of 2 weeks.

DETAILED DESCRIPTION:
Effective and safe methods are required to achieve substantial and long-lasting weight-loss with minimal and preferably no impact on the non-morbid obese individuals' pre-procedure lifestyle. The current available treatments for obesity in general and non-morbid obesity in particular, are, for the most part, ineffective in the long run and are associated with material adverse events and potentially lethal complications.

Sensate™, is an endoscopically-delivered, inner-stomach-wall-anchored, low-profile device (practically the exact size and shape of the famous Given Imaging PillCam™ swallowable device), which is advantageous in comparison to both open and minimally invasive surgical methods for treating obesity. The reason for that is because of the simple endoscopic delivery, inner-antrum-wall-anchoring and removal procedures are safe, minimally-invasive, requiring minimal participant sedation (not deep anesthesia), not requiring unique gastroenterologist skills, and can be done in an outpatient clinic setting just like in the hospital setting. Moreover, Sensate™ is designed to modestly reduce food consumption concurrently with the generation of greater satiety, and thus maintain balanced and healthier weight loss over a long period of time without mandating complementary radical lifestyle changes and nutritional changes which have been proven to be very hard and impractical on the obese individual.

This study will be the first study in humans, and it is focused on examining and validating the safety, tolerability and preliminary efficacy of Sensate™ in humans.

The Sensate™ study is comprised of two sequential cohorts of generally healthy patients with non-morbid obesity, with two participants in the first cohort and eight subjects in the second cohort. The first cohort is starting with just 2 subjects, in order to validate the absolute safety of the device and its delivery before additional subjects are being recruited. The sample size is the minimal one required to collect safety, tolerability and preliminary efficacy data. Participants will undergo screening to determine their health status and their eligibility to participate in the study. Screening examinations include medical history, physical examination, vital signs, weight measurement and laboratory assessments. Eligible patients will undergo an endoscopic device delivery procedure during which the device will be anchored in the inner stomach wall at the distal anterior antrum. Patients will be requested to complete a detail daily diary based on visual analogue scale (VAS) to record their eating sensations during and after each meal throughout the study. Physical examination, recording of adverse events and weight measurements will be conducted on day 14 and 28. In addition, phone calls are made every week during the study period to ask the patient about any health alterations. Endoscopic safety evaluation to validate that the device is anchored properly with no safety issues will be performed on Days 14 and 28 in the first two subjects and at day 28 for the remaining eight subjects. The device and its anchor will be completely removed endoscopically after 8 weeks. The participants will be followed-up for safety evaluation for an additional period of 2 weeks. Safety evaluations include physical examination, vital signs, adverse events and laboratory assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, 25 years of age or older and 55 years of age or younger at the time of the first screening visit.
* BMI (Body Mass Index) prior to the first screening visit between 35 - 40 kg/m2.
* General good health confirmed by medical history, physical examination, medication use in the 30 days prior to the baseline visit, and clinical chemistry and hematology lab test results.
* For women of childbearing potential: negative pregnancy test and willingness to use effective contraception during the entire study period.
* Signed informed consent to participate in the study.
* Ability of the participant to comply with all the requirements of the study and participate in all the intensive activities of the study throughout the study period.

Exclusion Criteria:

* Any contraindication to undergoing endoscopic and/or laparoscopic procedures.
* Known gastric motility disorder and/or history of chronic constipation problems.
* Known peptic ulcer and/or previous gastrointestinal antrum and/or pyloric surgery (open or laparoscopic) and/or structural abnormalities of the gastrointestinal tract (drop out criteria).
* History of chronic intestinal diseases or disorders.
* Prior obesity prevention surgical procedure (intra-gastric balloon, Lap band™ procedure, Bariatric surgery or others).
* Significant weight fluctuations (greater than ±5 kg) within the period of three months prior to first screening visit.
* Participants with significant eating pattern alterations according to participant interview.
* Current systemic intake of laxatives, steroids, non-steroidal anti-inflammatory medications, anticoagulants within 30 days prior to the screening visit and for the entire study duration.
* Participants who have a clinically significant or unstable medical or surgical condition that may preclude safe and complete study participation. Such conditions include significant gastrointestinal, cardiovascular, vascular disease, pulmonary/respiratory, hepatic impairment, renal, metabolic diseases, endocrinological, neurological, immune-deficiency, hematopoietic disease, or malignancies as determined by medical history, physical examination, or laboratory tests.
* Participants with any clinically significant abnormality upon physical examination or in the clinical laboratory test values such as abnormal blood test or abnormal blood coagulation test results prior to the baseline visit.
* Participants with any acute medical situation (e.g. severe febrile illness) or any uncontrollable infection, which is considered of significant by the Principal Investigator.
* Participants who have participated in another clinical trial of any kind within three months prior to the screening visit.
* Organ allograft.
* For female participants: planned pregnancy within 6 months from study start, active pregnancy, or breast-feeding.
* For male participants: intention to have a child within 6 months from the baseline visit.
* Any form of substance abuse (including drug or alcohol abuse), psychiatric disorder, or any chronic condition susceptible, in the opinion of the investigator, of interfering with the conduct of the study.
* Participants who are likely to be non-compliant or uncooperative during the study.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2008-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Adverse Events (subjective participant reporting or documentation). | 12 weeks

SECONDARY OUTCOMES:
Vital signs. Laboratory tests. Pathological findings in physical Examination and in endoscopic examination of stomach. Concomitant medication use. Body weight measurements. Improved VAS-based score. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Kiesslich, Univ.-Prof. Dr. med., Principal Investigator — Johannes Gutenberg University Mainz, I. Med. Klinik und Poliklinik
Locations (1):
- Johannes Gutenberg University, I. Med. Klinik, Mainz, Rhineland-Palatinate, Germany